CLINICAL TRIAL: NCT00147472
Title: A Prospective Cohort Study to Determine the Sensitivity of Positron Emission Tomography (PET) in Detecting Metastatic Cancer in Neck Lymph Nodes in Patients With Squamous Cell Head & Neck Cancer Managed With Primary Radiation Therapy
Brief Title: Positronic Emission Tomography (PET) Imaging in Post Radiation Evaluation of Head and Neck Tumours (PET PREVENT Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTA-Control-088421
Record Dates: First submitted 2005-09-01; First posted 2005-09-07 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Cancer of the Head and Neck
Keywords: Head and neck; Cancer; Diagnosis; Fluorodeoxyglucose; Positron-Emission Tomography; PET; Oncology
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET (Other): All patients receive PET scan and conventional CT imaging.
  Interventions: Other: PET scan in addition to conventional CT imaging

INTERVENTIONS:
Other: PET scan in addition to conventional CT imaging — PET scans, Pre and post radiation treatment
  Other Names: FDG PET

SUMMARY:
The purpose of this trial is to determine the ability of positron emission tomography (PET) to detect residual cancer in neck lymph nodes of patients following curative treatment with radiation therapy for squamous cell cancer arising in the head and neck.

Patients with head and neck cancer (HNC) undergo treatment of curative intent; patients who are node positive (N2 N3 stages) undergo standard management which includes post-radiation planned neck dissection but two thirds of patients end up not having evidence of residual disease in neck dissection specimens; these patients could have avoided surgery. However, currently used standard tests, like computed tomography (CT) and/or magnetic resonance imaging (MRI) cannot reliably predict who is post-radiation disease free.

DETAILED DESCRIPTION:
PET-Fluorodeoxyglucose scanning is an imaging test based on the increased uptake of radiolabelled glucose by tumour cells. PET might detect neck tumours better than other imaging tests. This is a cohort study in which patients with N2 N3 squamous cell carcinoma of the head and neck undergo a PET and a CT scan at baseline and then post-radiation therapy and chemotherapy. Then, they undergo neck dissection surgery. The PET and CT results are compared with the presence or absence of tumours in the neck nodes. If PET is sufficiently accurate in predicting the presence or absence of tumours in the neck nodes, then a neck dissection could be avoided.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be satisfied:

1. Histological evidence of squamous cell carcinoma of the head & neck (T1-T4 arising in either the oral cavity, larynx & pharynx, except Nasopharyngeal carcinoma);OR patients with histological evidence of squamous cell carcinoma metastatic to the neck and an unknown primary site after conventional workup without any of the following: i). Clinically suspected skin primary or previous diagnosis of skin cancer arising in the head and neck area; ii). Patients of Asian or African decent -possible nasopharynx primary; iii). Patients whose malignant adenopathy is confined to zone V -possible nasopharynx primary; and iv). Patients whose malignant adenopathy is confined to zone IV (supraclavicular)-possible lung primary.
2. Presence of advanced N2 or N3 neck disease.
3. Planned for primary curative radiation therapy (± chemotherapy) followed by neck dissection eight to twelve weeks after completion of treatment.

Exclusion Criteria:

1. Presence of distant metastasis
2. Recurrent tumour
3. Prior neo-adjuvant chemotherapy
4. Previous radiation therapy to intended treatment volumes
5. Other active malignancy
6. Surgically inoperable neck disease
7. Unable to remain supine for 60 minutes
8. Unfit to undergo general anesthetic or neck dissection for medical reasons
9. Known hypersensitivity to CT contrast
10. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-05; Primary Completion 2009-08 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Ability of PET compared to CT in identifying the presence of tumour in neck nodes | 2 years

SECONDARY OUTCOMES:
Tumour at the primary site 8-10 weeks following radiation; | 2 years
The change in PET signal (standard uptake value; | 2 years
Local recurrence, distant metastases and survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Waldron, MD, Study Chair — Princess Margaret Hospital, Canada; Ralph Gilbert, MD, Principal Investigator — Princess Margaret Hospital, Canada; Libni Eapen, MD, Principal Investigator — Ottawa Regional Cancer Centre; Anne Keller, MD, Principal Investigator — Princess Margaret Hospital, Canada; Mark N Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); Bayardo Perez-Ordonez, MD, Principal Investigator — Princess Margaret Hospital, Canada; Chu-Shu Gu, M.Sc., Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (4):
- Canada (4):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario